CLINICAL TRIAL: NCT02433704
Title: Preoperative Antibiotic Dosing for Total Knee Arthroplasty: Intraosseous Versus Systemic Infusion
Brief Title: Preoperative Antibiotic Dosing for Total Knee Arthroplasty
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty with enrollment
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00061712
Record Dates: First submitted 2015-04-10; First posted 2015-05-05 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2015-11

CONDITIONS: Acute Infection of Total Knee Replacement
MeSH Terms: interventions — Cefazolin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intraosseous Administration (Active Comparator): Cefazolin 1 gram will be given through an intraosseous cannula, placed into the medial aspect of the proximal tibia, after draping and before skin incision. The cefazolin will be administered as a bolus in 200 mL of normal saline.
  Interventions: Device: New Intraosseous; Drug: Cefazolin
- Systemic Intravenous Administration (No Intervention): Historical controls will be used and will have received systemic dosing of cefazolin within one hour of the incision.

INTERVENTIONS:
Device: New Intraosseous — Intraosseous administration of prophylactic antibiotics
  Arms: Intraosseous Administration
Drug: Cefazolin — Cefazolin 1 gram will be given through an intraosseous cannula, placed into the medial aspect of the proximal tibia, after draping and before skin incision. The cefazolin will be administered as a bolus in 200 mL of normal saline.
  Arms: Intraosseous Administration

SUMMARY:
To directly compare acute infection rates in patients undergoing total knee replacement with intraosseous regional administration or systemic intravenous administration of prophylactic antibiotics.

DETAILED DESCRIPTION:
Subjects will be prospectively enrolled into the Intraosseous Regional Administration (IORA) group, and the investigators will use historical controls for the Systemic Intravenous Administration (SIA) group, to include a matched group of patients from 6 months prior to enrollment. SIA group will receive systemic dosing of cefazolin within one hour of the incision, which is the current standard of care. IORA group will receive intraosseous dosing after the tourniquet is inflated to 300-350mm/Hg. Cefazolin 1 gram will be given through an intraosseous cannula, placed into the medial aspect of the proximal tibia, after draping and before skin incision. The cefazolin will be administered as a bolus in 200 mL of normal saline. Incision will be made immediately after infusion. Subjects in both groups will receive routine care following the procedure. Primary outcome will be acute surgical site infection, which is defined as within 3 weeks after the surgical procedure. Secondary outcomes will include correlation of clinical comorbidities to the primary outcome, report complications, and compare surgery specific information (tourniquet time, blood loss).

Subjects with a penicillin allergy will receive a 200mg cefazolin test dose via a systemic intravenous route, which is the current standard of care. If no adverse reaction is observed, then the investigators will proceed with administration of 1g cefazolin via the intraosseus route.

ELIGIBILITY:
Inclusion Criteria:

•primary diagnoses of osteoarthritis

Exclusion Criteria:

* history of compartment syndrome
* allergy to an antibiotic in the study
* venous stasis
* peripheral vascular disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
rate of acute surgical site infection | defined as within 3 weeks after the surgical procedure

SECONDARY OUTCOMES:
correlation of clinical comorbidities to acute infection rates | 1 year post surgical intervention
number of complications | 1 year post surgical intervention
tourniquet time | during procedure, up to approximately 2.5 hours
blood loss | during procedure, up to approximately 2.5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Wellman, MD, Principal Investigator — Duke University
Locations (1):
- Duke Medical Plaza Page Road, Durham, North Carolina, United States